CLINICAL TRIAL: NCT05664451
Title: Improving Nonsurgical Treatment of Urinary Incontinence Among Women in Primary Care in Wisconsin: Bridging Community-based Continence Promotion and Primary Care
Brief Title: WI-INTUIT: Bridging Community Based Continence Promotion and Primary Care
Acronym: WI-INTUIT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: MetaStar, Inc. (Industry); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kathryn Flynn, Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021-1477; PRO00042157 (Other: Medical College of Wisconsin); 1U18HS028738-01 (AHRQ)
Record Dates: First submitted 2022-11-07; First posted 2022-12-23 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Streamlined Practice Facilitation (SPF) implementation of UI-Assist (Active Comparator): Streamlined practice facilitation encompasses multiple well-established strategies from the Expert Recommendations for Implementing Change (ERIC) as field-tested in and updated after EvidenceNOW. To ensure the interventions and tools offered are consistent across practices, practice facilitators will receive training and support on UI-Assist, milestones, tracking tools for documenting changes made by sites, etc. according to a Practice Facilitation Training Manual and toolkit that will be built based on ones used for prior EvidenceNOW initiatives.
  Interventions: Behavioral: UI-Assist
- Streamlined Practice Facilitation (SPF) + Partnership Building (PB) implementation of UI-Assist (Experimental): In addition to streamlined practice facilitation, those practices allocated to Streamlined Practice Facilitation plus Partnership Building (SPF+PB) will have facilitation and configurable solutions that engage community resources and enable coalition building. In addition to a MetaStar practice facilitator, a partnership facilitator from the Wisconsin Institute for Healthy Aging (WIHA) will identify existing local community resources with which the practice may choose to partner.
  Interventions: Behavioral: UI-Assist; Other: Partnership Building

INTERVENTIONS:
Behavioral: UI-Assist — To support primary care in implementing guideline-based care, it is helpful to distill interventions to their key components, such as the five major intervention steps for tobacco use and dependence (the "5 A's"). The 5 A's (Ask, Advise, Assess, Assist, Arrange) has been shown to help primary care providers implement clinical practice guidelines with minimal additional burden. The 5 A's can be similarly simplified for urinary incontinence (UI) screening and treatment to Ask (screen for UI); Advise (inform that effective nonsurgical treatments exist); and Assist (help patient get treatment with pharmacotherapy, referral to community classes, physiotherapy or urology / urogynecology).
Other: Partnership Building — In addition to the strategies described above, those practices allocated to streamlined practice facilitation and partnership building will have facilitation and configurable solutions that engage community resources and enable coalition building. In addition to a practice facilitator, a partnership facilitator from the Wisconsin Institute for Healthy Aging (WIHA) will identify existing local community resources with which the practice may choose to partner. After initiating academic detailing, these practices will have further access to Drs. Brown and Neuner for ongoing consultation. An online learning community will also be created where information can be shared and exchanged throughout the duration of the project and beyond the maintenance phase.
  Arms: Streamlined Practice Facilitation (SPF) + Partnership Building (PB) implementation of UI-Assist

SUMMARY:
This project seeks to determine whether primary care practices that receive supplemental partnership building implement UI-Assist with higher fidelity than practices that receive streamlined practice facilitation alone.

DETAILED DESCRIPTION:
This quality improvement research project is one of five across the country funded by the Agency for Healthcare Research and Quality (AHRQ) through the EvidenceNOW Managing Urinary Incontinence initiative titled: "Improving Nonsurgical Treatment of Urinary Incontinence among women in Primary Care." The purpose of this national initiative is to identify implementation strategies that best support primary care practices in delivering high quality care for urinary incontinence. Components of high-quality care including screening, diagnosing, and offering non-surgical first-line treatments for urinary incontinence in women, all of which already occur in primary care.

The WI-INTUIT quality improvement project compares two implementation strategies to implement UI-Assist, an intervention to support primary care practices in increasing their rates of screening, diagnosing, and treating urinary incontinence in their adult female patients: (1) streamlined practice facilitation (SPF) and (2) streamlined practice facilitation in combination with partnership building (SPF+PB).

ELIGIBILITY:
This is an organizational intervention. Outcomes will be evaluated at the population-level by facility.

Primary Care practices in Wisconsin serving female adults:

Inclusion Criteria:

* Patients must be 18 years or older and be assigned female at birth
* Practices must have and be willing to provide key data from electronic health records
* Practices willing to participate in partnership building activities (randomly allocated)
* Practices willing to work with a practice facilitator to implement UI-Assist in their practice

Exclusion Criteria:

- No additional exclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients are eligible to participate in this study if they were assigned female at birth.
Enrollment: 40 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Differences in Screening Rates for Urinary Incontinence | 3 months, 10 months
  Defined as the rate of eligible patients screened for urinary incontinence (UI) at preventive visits. Data on UI screening and patient eligibility will be ascertained through responses to a short post-visit patient survey. Patients will be asked five questions to determine if their healthcare team screened for and, if necessary, provided them with treatment options for UI. Preventive visits include visits classified as: a preventive visit, a physical exam, or a Medicare annual wellness visit.

SECONDARY OUTCOMES:
Differences in scores on Patient-Reported Outcomes Measurement Information System (PROMIS) - Global Health | 10 months, 13 months
  This 10-item survey measures symptoms, functioning, and quality-of-life for various chronic conditions and diseases. Two overall scores are calculated: a Global Physical Health Score and a Global Mental Health Score. Response options are on a 5-pt scale. Each score has a range of 0-20, 0 represents most severe mental and physical impairment, 20 represents the best state of health possible.
Differences in bowel leakage symptoms | 10 months, 13 months
  This 4-item survey assesses patient experience with accidental bowel leakage in terms of frequency (Rarely, Sometimes, Weekly, Daily, I don't know), amount of leakage (Gas only, Small amount of stool, Moderate amount of stool, Large bowel movement, I don't know) and seeking care (Yes, No, I don't know).
Differences in scores on Patient-Reported Outcomes Measurement Information System (PROMIS) - Constipation | 10 months, 13 months
  This 3-item scale measures patient's difficulty with passing bowel movements within the past 7 days. Question responses are Never, One day, 2-6 days, Once a day, More than once a day or Never, Rarely, Sometimes, Often, Always. Higher scores indicate patients have a greater difficulty with passing bowel movements.
Self-reported changes: changes in usage of urinary incontinence coping strategies | 10 months, 13 months
  This item ascertains whether the individual has tried to use any urinary incontinence coping strategies "Have you tried any strategies to improve your urinary incontinence/ leakage?" Response options: "Yes, No, I don't know". The uptake in strategies between baseline and 90-day follow-up will be assessed.
Self-reported changes: change in money-spent on incontinence treatments | 10 months, 13 months
  Self-reported changes: change in out-of-pocket costs of incontinence treatments to manage symptoms. This will be ascertained by asking participants how much money have they spent on products to manage their symptoms.
Self-reported changes: urinary incontinence treatments adopted | 10 months, 13 months
  This item addresses which urinary incontinence treatment strategies the individual implemented "If yes, what strategies did you try? Please select all that apply." Response options: (1) Making changes to what you eat or drink; (2) Making changes to how often you urinate; (3) Wearing pads, panty liners, or disposable undergarments (diapers); (4) Doing pelvic floor muscle exercises (Kegels) on your own; (5) Doing pelvic floor muscle exercises (Kegels) with a therapist; (6) Using a medication; (7) Stopping a medication; (8) Using a pessary (something that sits inside the vagina to help with urine leakage); (9) Having a procedure (for example, injections to the bladder, electrical stimulation, or surgery); (10) Something else: ______
Self-reported changes: change in pad use | 10 months, 13 months
  Self-reported changes: change in the number and type of pad(s) used
Global perception of improvement (GPI) | 13 months
  Global perception of improvement (GPI) is a tool for Global Rating of Patient Satisfaction and Perceptions of Improvement.
  This item asks patients if they feel their urinary incontinence has changed over the past 90 days. Participants are able to select one of the following options: very much better, much better, a little better, no change, a little worse, much worse, very much worse.
Practice contextual factors - reach | 1 month
  This questionnaire collects practice-level demographic information including: setting, general patient demographic information, general provider-level information, practice patterns, and relationships with other health care systems.
Difference in scores of the Change Process Capability Questionnaire (CPCQ) Strategies Scale | 1 month, 9 months
  This validated instrument assesses practice systems ability to implement change by measuring attitudes and experience with implementation strategies in a Likert rating scale.
  Each response to the CPCQ survey is coded so that 2=strongly positive, 1=positive, 0=neutral, -1=negative, and -2=strongly negative. The coded responses are summed to create a strategies score, with the score ranging from -28 to +28. More negative scores are associated with lower use of strategies and more positive scores are associated with higher use of strategies.
Organizational Readiness for Implementing Change | 1 month, 9 months
  This 12-item survey measures how well employees at an organization feel they can implement the change in processes proposed by an intervention. Each of the 12-items is measured by a Likert scale (1=Disagree through 5=Agree). Responses are summed; higher scores indicate participants are more likely to initiate change, exert greater effort, and exhibit greater persistence; whereas, lower scores indicate the opposite.
Clinical Staff Questionnaire in the National Demonstration Project - Community knowledge | 1 month, 9 months
  The community knowledge subset of the Clinical Staff Questionnaire, consists of four questions on a Likert scale (1=strongly disagree, 2=disagree, 3=neutral, 4=agree, 5=strongly agree). Scores on this subset will be summed and then averaged for each individual's response (score range: 1 to 5). Items will be reverse-scored when appropriate so that higher numbers reflect more positive ratings.
Clinical Staff Questionnaire in the National Demonstration Project - Practice adaptive reserve | 1 month, 9 months
  The practice adaptive reserve subset of the Clinical Staff Questionnaire, consists of 23 questions on a Likert scale (1=strongly disagree, 2=disagree, 3=neutral, 4=agree, 5=strongly agree). Scores on this subset will be summed and then averaged for each individual's response (score range: 1 to 5). Items will be reverse-scored when appropriate so that higher numbers reflect practices' ability to make and sustain change.
Change in response to a single-item burnout measure | 1 month, 9 months
  The single-item burnout measure, adapted from the Mini Z Burnout survey, assesses healthcare staff burnout. Responses are 1-5, with scores of 3 or higher defining high burnout.
Change in response to Urinary Incontinence Assist Project Practice Survey | 6 months, 9 months, and 12 months
  All clinic staff members will be asked about their experience implementing the UI-Assist tool. The survey will ask individuals to rate various aspects of their clinic's prior experiences with urinary incontinence on a Likert scale (Not at all, slightly, somewhat, very, extremely). Individuals will be asked questions pertaining to the ease of incorporating UI-Assist into their project on a Likert scale, as well as questions pertaining to the perception of the project in their clinic on a Likert scale (1=strongly disagree through 7=strongly agree).
Differences in scores of the International Consultation on Incontinence Questionnaire-Urinary Incontinence (ICIQ-UI) | 10 months, 13 months
  ICIQ-UI is a subjective measure of severity of urinary loss and quality of life for those with urinary incontinence. It is scored on a scale from 0-21. Based on the score participant can be placed in four severity categories: slight (1-5), moderate (6-12), severe (13-18) and very severe (19-21).
Differences in scores of Incontinence Impact Questionnaire (IIQ-7) | 10 months, 13 months
  The Incontinence Impact Questionnaire - Short Form (IIQ-7) will be used to assess areas in a patient's life that may have been influenced or changed by their urinary incontinence. Patients are asked to select the response that best describes how much their activities, relationships, and feelings are being affected by urinary incontinence. Item responses are assigned values of 0 for "not at all," 1 for "slightly," 2 for "moderately," and 3 for "greatly." The average score of items responded to is calculated. The average, which ranges from 0 to 3, is multiplied by 33 1/3 to put scores on a scale of 0 to 100. A score <50 indicates good quality of life, between 50-70 indicates moderate quality of life, and >70 indicates poor quality of life.
Patients' health literacy level | 10 months
  Patients will be asked four questions to determine their health literacy level through the BRIEF - health literacy screening tool. Each item is worth 1 to 5 points depending on their response. Add the values for the four responses to get a total score, which can range from a minimum of 4 to a maximum to 20. A score of 4 - 12 (limited) indicates the patient is not able to read most low literacy health materials; will need repeated oral instructions; materials should be composed of illustrations or video tapes. Will need low literacy materials; may not be able to read a prescription label. A score of 13 - 16 (marginal) indicates the patient may need assistance; may struggle with patient education materials. A score of 17 - 20 (adequate) indicates the patient will be able to read and comprehend most patient education materials.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Neuner, MD, MPH, Principal Investigator — Medical College of Wisconsin
Locations (3):
- United States (3):
  - Kaiser Permanente, San Diego, California
  - MetaStar, Inc., Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel UJ, Moureau MK, Neuner JM, Brown HW. Screening and Treating Urinary Incontinence in Primary Care: A Missed Opportunity. OBM Geriat. 2023;7(4):252. doi: 10.21926/obm.geriatr.2304252. Epub 2023 Oct 5. PMID 38567050